CLINICAL TRIAL: NCT06117397
Title: A Text Messaging Intervention to Reduce Perinatal Depression Risk
Acronym: PTMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Yale University (Other); Michigan State University (Other); Worcester Polytechnic Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kimberly A. Yonkers, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 00000462; R34MH130934-03 (NIH)
Record Dates: First submitted 2023-05-01; First posted 2023-11-07 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Episode

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text4Moms (Experimental): Texts will include video links that reinforce information relevant to Interpersonal Psychotherapy (IPT).
  Interventions: Other: Text Messaging Intervention
- Educational Control (No Intervention): The control condition will be limited to texts related to pregnancy, nutrition and sleep. We will avoid elements that have behavioral therapeutic effects. Although this condition is meant to constitute time and attention control, we will include material on recognizing depression and links to ways to attain depression treatment and suicide hotline information.

INTERVENTIONS:
Other: Text Messaging Intervention — A text messaging intervention that includes enhanced content such as tailoring, video links and a chat function
  Arms: Text4Moms

SUMMARY:
Development and preliminary testing of a text messaging intervention that will reduce the risk of a major depressive episode and worsening depressive symptoms in perinatal individuals. The system will screen pregnant individuals, send tailored text messages with links to enhanced content, and will include a peer chat function.This accessible text platform will leverage both the ease of use inherent in text messages and the power of enhanced content drawn evidence from based behavioral interventions (Interpersonal Therapy).

DETAILED DESCRIPTION:
About 1 in 7 pregnant individuals experience depression, with roughly the same number facing this devastating illness after delivery. The downstream effects of perinatal depression adds to its toll with increased risk of preterm birth; impairments in maternal-child attachment; adverse effects on infant development; and decreased breastfeeding initiation/duration. The US Preventative Services Task Force finds that some major depressive episodes (MDEs) can be averted with counseling strategies that employ principles from interpersonal therapy (IPT). They also observe the value of peer support, which can decrease perinatal depression. A possible shared mechanism for these interventions is enhancement of self-efficacy, which is critical in the setting of stressful events such as pregnancy and parenting. However, practical implementation of interventions to reduce depression risk is challenging. Reproductive health providers have limited time and training to deliver depression prevention programs. As well, perinatal individuals may not appreciate the need to participate in a prevention program or have difficulty finding or affording providers of behavioral interventions. Technology can assist with these challenges by providing education, support and therapeutic interventions to perinatal individuals. Unlike web-based applications (apps), text messaging interventions (TMIs) can proactively deliver health information and messages, even to those with limited motivation to engage in preventative interventions. Mobile phone use has exploded with >95% of pregnant individuals (including >85% of the minority population) reporting use of a mobile phone to communicate via short text messages. TMIs can also screen perinatal individuals for depression outside the general medical setting and provide general peer support. With end-user input throughout the process, the investigators will build a multi-component TMI (called Text4Moms) that screens and triages perinatal individuals for risk of a MDE. This system will draw content from IPT; it will send tailored text messages with links to relevant video content to perinatal individuals at risk for a depressive episode. An on-demand secure chat function staffed by a peer with lived experience will complement the text messages for enhanced support. The system will include pre-populated content for peers to cut and paste into text messages for participants, which will support peers and decrease their training burden. This system leverages some of the best components of an app (video, tailoring, chat) into a common and user-friendly text messaging platform. After development, the investigators will conduct a pilot randomized trial to test the ability of the TMI to enhance the target of self-efficacy and decrease depressive symptoms and risk of a MDE. The investigators will query Research Domain Criteria (RDOC) constructs of "loss" and "threat," and will evaluate preliminary effectiveness and implementation (assessment of feasibility, acceptability, use and benefit of the peer chat feature) through a pilot randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* "At risk" as determined by an Edinburgh Postnatal Depression Scale score of at least 9, or an average score >3 on the 6-item Medical Outcomes Social Support Survey or history of depression in pregnancy or postpartum depression
* At least age 16
* Are willing and able to provide informed consent
* Are willing to use a smart phone to receive texts

Exclusion Criteria:

* In a major depressive episode
* Planning on terminating pregnancy
* Have panic disorder or substance use disorder
* Currently in behavioral health care treatment
* Blind individuals
* Permanently living in an institutional setting

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Edinburgh Prenatal Depression Scale | Week 4 for pre-pilot and week 8 for pilot, adjusted for baseline
  10-item continuous measure of depression. Self-report that will be administered by computer. Will be administered three times (for pre-pilot administered at screening, 2 weeks, and 4 weeks; for pilot administered at screening, 4 weeks, and 8 weeks). Items are scored 0-3, with a maximum score of 30. Higher scores show increased severity.
General Self Efficacy Scale | Week 4 for pre-pilot and week 8 for pilot, adjusted for baseline
  10 item measure of self efficacy. Items are scored 1-4, with scores ranging between 10 and 40. A higher score indicates more self-efficacy. Will be administered three times (for pre-pilot administered at baseline, 2 weeks, and 4 weeks; for pilot administered at baseline, 4 weeks, and 8 weeks).
System Usability Scale | Week 4 for pre-pilot and week 8 for pilot, adjusted for baseline
  10 items rated on a 1-5 scale, with scores ranging from 0-100, with a higher score indicating greater acceptability. Will be administered one times (for pre-pilot administered at 4 weeks; for pilot administered at 8 weeks).
Patient engagement with text messages | 0-8 weeks
  Percentage of participants opening >80% of text messages and clicking on >30% of links to enhanced content.
Patient engagement with chat | 0-8 weeks
  Percentage of participants engaging with chat and endorsing 4 out of 5 on its utility.

SECONDARY OUTCOMES:
Diagnosis of a major depressive episode | Week 4 for pre-pilot and week 8 for pilot, adjusted for baseline
  Diagnosis of a major depressive episode using the PHQ-9, the Major Depressive Disorder module of the full PHQ. Will be administered three times (for pre-pilot administered at screening, 2 weeks, and 4 weeks; for pilot administered at screening, 4 weeks, and 8 weeks).
User Engagement Scale | Week 4 for pre-pilot and week 8 for pilot, adjusted for baseline
  12 items rated on a 1-5 scale, with scores ranging from 10-50, with higher scores indicating greater acceptability, with an average score of 80.3. Will be administered one time (for pre-pilot administered at 4 weeks; for pilot administered at 8 weeks).
Perlin Mastery Scale | Week 4 for pre-pilot and week 8 for pilot, adjusted for baseline
  7 items scaled on a 1-4 scale, with scores ranging from 7-28. Low scores indicate low mastery. Will be administered one time at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Yonkers, MD, Principal Investigator — UMass Chan Medical School
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We welcome any interest in using or modifying the intervention materials developed under this project, which will be aided by our use of the Computerized Intervention Authoring System (CIAS) platform. Our overall plan will include presentations at national scientific meetings as well as publication of results, via reputable peer-reviewed journals and the National Library of Medicine/PubMed Central. We will deposit this dataset with the National Database for Clinical Trials Related to Mental Illness. We will indicate in publications and presentations where and how to access these data. Study materials and information regarding access to intervention content will be made available via the Open Science Framework (OSF).
  Individuals who would like our data can also complete a "data analysis requisition form" that describes their specific hypotheses with mock-ups of tables. All data will be de-identified before sharing. We will make the data available under a data sharing agreement.
Supporting Information: Study Protocol, SAP
Time Frame: 12 months after data analysis
Access Criteria: interest in postpartum depression

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/97/NCT06117397/Prot_SAP_000.pdf